CLINICAL TRIAL: NCT01528215
Title: An Open, Prospective, Randomized, Multicenter Study Comparing OsseoSpeed™ EV With OsseoSpeed™ TX in Partially Edentulous Maxillae and Mandibles. A 5-year Follow-up Study.
Brief Title: Multicenter Study Comparing OsseoSpeed TX With OsseoSpeed EV.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTX-PLUS-0001
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Partial Edentulism in the Maxilla or in the Mandible

ARMS (2):
- OsseoSpeed EV (Experimental): OsseoSpeed EV implants; Ø 3.6, 4.2, 4.8 mm in lengths of 9,11 and 13 mm
  Interventions: Device: OsseoSpeed EV
- OsseoSpeed TX (Active Comparator): OsseoSpeed TX implants; Ø 3.5, 4.0 and 5.0 mm in lengths of 9,11 and 13 mm
  Interventions: Device: OsseoSpeed TX

INTERVENTIONS:
Device: OsseoSpeed EV — OsseoSpeed EV implants; Ø 3.6, 4.2, 4.8 mm in lengths of 9,11 and 13 mm
  Arms: OsseoSpeed EV
Device: OsseoSpeed TX — OsseoSpeed TX implants; Ø 3.5, 4.0 and 5.0 mm in lengths of 9,11 and 13 mm
  Arms: OsseoSpeed TX

SUMMARY:
The purpose of this study is to evaluate the outcome of implant OsseoSpeed EV compared to implant OsseoSpeed TX with regards to marginal bone level changes and implant survival rate up to five years after implant loading. The hypothesis is that there will be no clinically relevant differences in marginal bone level alterations one year after functional loading.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of Informed Consent.
2. 18 -75 years at enrollment.
3. In need of implant(s) replacing missing tooth/teeth in the maxilla or in the mandible (no edentulous jaws).
4. History of edentulism in the planned implant area of at least 3 months (at Visit 2).
5. At least 4 months of healing after last grafting procedure in the planned implant area (at Visit 2).
6. Deemed by the investigator to be suitable for one stage surgery and be likely to present an initially stable implant situation i.e. have a bone height and bone width suitable for the chosen study implants.
7. Deemed by the investigator to be suitable for loading after 6-8 weeks.
8. Deemed by the investigator to have a "functional" opposing dentition at the time of loading the implants i.e. an even distribution of contacts between the teeth in the opposite jaw and the planned permanent crown/bridge.

Exclusion Criteria:

1. Unlikely to be able to comply with study procedures, as judged by the investigator.
2. Uncontrolled pathological processes in the oral cavity.
3. Untreated, uncontrolled caries and/or periodontal disease.
4. Known or suspected current malignancy.
5. History of radiation therapy in the head and neck region.
6. History of chemotherapy within 5 years prior to surgery.
7. Systemic or local disease or condition that would compromise post-operative healing and/or osseointegration, as deemed by the investigator.
8. Uncontrolled diabetes mellitus.
9. Corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration.
10. Smoking more than 10 cigarettes per day.
11. Present alcohol and/or drug abuse.
12. Current need for bone grafting and/or augmentation in the planned implant area. Local, minor soft tissue grafting will be allowed.
13. Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site).
14. Previous enrollment in the present study.
15. Simultaneous participation in other clinical studies at enrollment (Visit 1) and during the subject's first year of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clark M Stanford, Prof, Principal Investigator — University of Illinois at Chicago, College of Dentistry
Locations (4):
- Dows Institute for Dental Research, University of Iowa, College of Dentistry, Iowa City, Iowa, United States
- University Hospital Ghent, Dental School Department Periodontology, Ghent, Belgium
- Dep. of Prosthodontics, Goethe University, Frankfurt am Main, Germany
- Dental private practice, Denis Cecchinato, Padua, Italy

REFERENCES:
- [Result] Stanford CM, Barwacz C, Raes S, De Bruyn H, Cecchinato D, Bittner N, Brandt J. Multicenter Clinical Randomized Controlled Trial Evaluation of an Implant System Designed for Enhanced Primary Stability. Int J Oral Maxillofac Implants. 2016 Jul-Aug;31(4):906-15. doi: 10.11607/jomi.4869. PMID 27447160

RESULTS

PARTICIPANT FLOW:
Period: Enrollment to 1 Year Follow-up
Arm/Group | OsseoSpeed EV | OsseoSpeed TX
Started | 59 | 61
Completed | 55 | 60
Not Completed | 4 | 1
Not completed — Adverse Event | 4 | 1
Period: 1 Year Follow-up to 5 Year Follow-up
Arm/Group | OsseoSpeed EV | OsseoSpeed TX
Started | 55 | 60
Completed | 40 | 45
Not Completed | 15 | 15
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 10 | 13
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OsseoSpeed EV | OsseoSpeed TX | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (16) | 51 (13) | 51 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 29 | 63
  Male | 25 | 32 | 57

OUTCOME MEASURES:

1. Primary Outcome: Marginal Bone Level Change After 1 Year in Use.
Description: Marginal bone level will be determined from radiographs and expressed as the distance from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal bone level expressed in millimeters at the 1 year follow-up visit compared to values obtained at delivery of permanent restoration i.e. loading (baseline). Positive value = bone gain, Negative value = bone loss.
Time Frame: Evaluated at implant loading and at the 1 year follow-up after implant loading.
Population: In the EV group, 55 subjects (73 implants) completed the 1 year follow-up visit.
  In the TX group, 60 subjects (84 implants) completed the 1 year follow-up visit. Three of the radiographs were not possible to evaluate, giving an overall number of 59 subjects (81 implants) as basis for the analysis of marginal bone level change.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed EV | OsseoSpeed TX
Number analyzed (Participants) | 55 | 59
Number analyzed (Implants) | 73 | 81
Millimeter | 0.27 (0.53) | 0.14 (0.47)

2. Secondary Outcome: Marginal Bone Level Change After 5 Years in Use.
Description: Marginal bone level will be determined from radiographs and expressed as the distance from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal bone level expressed in millimeters at the 5 years follow-up visit compared to values obtained at delivery of permanent restoration i.e. loading (baseline).
Time Frame: Evaluated from implant loading to the 5 years follow-up after implant loading.
Population: In the EV group, 40 subjects (52 implants) completed the 5-year follow-up visit.
  In the TX group, 45 subjects (64 implants) completed the 5-year follow-up visit.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed EV | OsseoSpeed TX
Number analyzed (Participants) | 40 | 45
Number analyzed (Implants) | 52 | 64
Millimeter | 0.24 (0.85) | 0.11 (0.85)

ADVERSE EVENTS:
Arm/Group | OsseoSpeed EV | OsseoSpeed TX
Serious Adverse Events (participants affected / at risk) | 13/59 | 13/61
Other Adverse Events (participants affected / at risk) | 0/59 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OsseoSpeed EV (N=59) | OsseoSpeed TX (N=61)
Colitis flare-up (Gastrointestinal disorders) | 1 | 0
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Infection causing swelling and difficulties swallowing (Infections and infestations) | 0 | 1
Prostate cancer (Renal and urinary disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Abdominal aortic aneurysm (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2
Breast cancer (Reproductive system and breast disorders) | 1 | 0
Onset of Diabetes (Endocrine disorders) | 1 | 3
Hip surgergy (Musculoskeletal and connective tissue disorders) | 1 | 0 — Hospitalisation due to surgery
Torn retina (Eye disorders) | 1 | 0
Cyst (Gastrointestinal disorders) | 1 | 0
Hernia neck (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer of oesophagus (Gastrointestinal disorders) | 1 | 0
Fibia fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Gastrointestinal disorders) | 0 | 1
High bloodpressure (General disorders) | 0 | 1
Insertion of cardiac stents (Cardiac disorders) | 0 | 1
Premature ventricular contractions (PVC) (Cardiac disorders) | 0 | 1
Death due to cerebral hemorrhage (Nervous system disorders) | 0 | 1
Thumb lost in accident (Musculoskeletal and connective tissue disorders) | 0 | 1
Aortic valve replacement surgery (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less